CLINICAL TRIAL: NCT05183243
Title: A Multicenter, Open-label Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics, and Preliminary Efficacy of GH21 Capsules in Subjects With Advanced Solid Tumors
Brief Title: GH21 Capsules for Advanced Solid Tumors: A Study on Safety and Early Results
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH21-CRS001
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor; Non-Small Cell Lung Cancer; Pancreatic Cancer; Colorectal Cancer; Head and Neck Neoplasm
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monotherapy Dose Escalation. (Experimental): Treatment with GH21 alone, conducted until disease progression, intolerance or end of study.
  Interventions: Drug: GH21 Capsule

INTERVENTIONS:
Drug: GH21 Capsule — GH21 for oral administration at doses of Dose A, Dose B, Dose C, Dose D, Dose E and Dose F.

SUMMARY:
Evaluate the safety and tolerability of GH21 in patients with advanced solid tumors.

Estimate the maximum tolerated dose (MTD) in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects greater than or equal to 18 years old；
2. Written informed consent obtained prior to any study-related procedure being performed;
3. Subjects with life expectancy ≥3 months;
4. Eastern Cooperative Oncology Group performance score 0 - 2;
5. Subjects must have histologically or cytologically confirmed advanced or metastatic solid tumor;
6. At least one measurable lesion based on RECIST version 1.1 .

Exclusion Criteria:

1. History of other malignancies within 3 years before screening,unless radical non-melanoma skin cancer or basal cell carcinoma of the skin or carcinoma in the situ of the cervix;
2. Have central nervous system metastases;
3. Prior treatment with SHP2 inhibitor;
4. Have major surgery within 28 days prior to the first dose of GH21;
5. Left ventricular ejection fraction (LVEF) <50 %;
6. Females who are pregnant or breastfeeding ;
7. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection;
8. Conditions that the investigator considers inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) of GH21. | 28 Days
  MTD is the highest dose of a treatment that does not cause unacceptable side effects.
Characterize the Safety of GH21 | Approximately 3 years
  Number of participants with treatment-emergent adverse events and serious AEs.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 3 years
  Based on assessment of radiographic imaging per RECIST version 1.1
Disease Control Rate (DCR) | Approximately 3 years
  Based on assessment of radiographic imaging per RECIST version 1.1
Duration of Response (DOR) | Approximately 3 years
  Based on assessment of radiographic imaging per RECIST version 1.1
Progression-Free Survival (PFS) | Approximately 3 years
  Based on assessment of radiographic imaging per RECIST version 1.1
PD of GH21 | Approximately 3 years
  Change of phosphorylated ERK
Cmax | Approximately 3 years
  The maximum or "peak" concentration of GH21 observed after administration
Tmax | Approximately 3 years
  The time to peak concentration of GH21
T1/2 | Approximately 3 years
  Half-life of GH21

CONTACTS AND LOCATIONS:
Overall Officials: Haidan Wang, Doctorate, Study Director — 0512-86861608
Locations (9):
- China (9):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Beijing University Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang

IPD SHARING:
Plan to Share IPD: No
NO plan